CLINICAL TRIAL: NCT03778229
Title: A Phase II Study Assessing the Efficacy of Osimertinib in Combination With Savolitinib in Patients With EGFRm+ and MET+, Locally Advanced or Metastatic Non Small Cell Lung Cancer Who Have Progressed Following Treatment With Osimertinib.
Brief Title: Osimertinib Plus Savolitinib in EGFRm+/MET+ NSCLC Following Prior Osimertinib
Acronym: SAVANNAH
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5084C00007; 2018-003012-51 (EudraCT Number)
Record Dates: First submitted 2018-11-30; First posted 2018-12-19 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma
Keywords: Non Small Cell Lung Cancer; epidermal growth factor receptor mutation positive; hepatocyte growth factor receptor; savolitinib; Osimertinib; AZD9291; AZD6094; volitinib
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — osimertinib; 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine

STUDY DESIGN:
Intervention Model Description: Under Protocol versions 1-6 the study model was single arm (open-label).
  Starting protocol version 7 patients will be randomised in a double blinded manner to receive savolitinib in combination with osimertinib or savolitinib with placebo to osimertinib with crossover option upon disease progression assessed by Investigator.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- osimertinib + savolitinib (Experimental): osimertinib + savolitinib
  Interventions: Drug: osimertinib; Drug: savolitinib
- placebo + savolitinib (Placebo Comparator): placebo + savolitinib
  Interventions: Drug: savolitinib; Drug: placebo

INTERVENTIONS:
Drug: osimertinib — osimertinib (80 mg oral OD).
  Arms: osimertinib + savolitinib
Drug: savolitinib — savolitinib (300 mg oral OD or 300 mg oral BID or 600 mg oral OD)
Drug: placebo — placebo to osimertinib (oral OD)
  Arms: placebo + savolitinib

SUMMARY:
This study (the SAVANNAH study) will investigate the efficacy of osimertinib in combination with savolitinib in patients with EGFRm+ and MET+, locally advanced or metastatic NSCLC who have progressed following treatment with osimertinib

DETAILED DESCRIPTION:
The combination of osimertinib with savolitinib in this study (the SAVANNAH study) will explore if the combination will overcome MET-amplification as a mechanism of resistance. The SAVANNAH study will investigate the efficacy of osimertinib in combination with savolitinib in patients with EGFRm+ and MET-amplified/overexpressed, locally advanced or metastatic NSCLC who have progressed following treatment with osimertinib.

Eligible patients will be those with histologically or cytologically confirmed diagnosis of EGFRm+, MET amplified/overexpressed (FISH10+ and/or IHC90+) NSCLC that is locally advanced or metastatic and is not amenable to further surgery or radiotherapy with curative intent. The disease must have progressed following treatment with first line osimertinib. Patients must have confirmation of MET-amplified/overexpressed tumour by central FISH and IHC testing (requirements summarised in the main body of the protocol and fully explained in the Central Laboratory Manual). Patients must not have received prior or current treatment with savolitinib or another MET inhibitor.

All patients confirmed as eligible will begin treatment on Day 1 with osimertinib + savolitinib combination therapy or placebo to osimertinib + savolitinib. Treatment will continue in 28 day cycles until either objective disease progression by investigator per RECIST 1.1 is assessed, unacceptable toxicity occurs, consent is withdrawn or another discontinuation criterion is met.

ELIGIBILITY:
Inclusion criteria:

* Patients must be ≥18 years of age (≥20 years of age in Japan). All genders are permitted.
* Histologically or cytologically confirmed locally advanced or metastatic EGFRm+ NSCLC harbouring an EGFR mutation known to be associated with EGFR TKI sensitivity and permitted in the osimertinib national label (such as either exon 19 deletion and/or L858R) which is not amenable to curative therapy.
* Documented radiologic disease progression on 1L osimertinib.
* MET amplification and/or overexpression (FISH10+ and/or IHC90+) as determined by FISH (central) and IHC (central) testing on tumour sample collected following progression on 1L osimertinib treatment.
* Available tumour sample for central MET FISH and IHC analysis or willingness to collect additional sample for central testing which fulfils the following requirements:

Obtained following progression on previous osimertinib therapy;

obtained within 2 years of submission for MET analysis;

sufficient tissue to meet the minimum tissue requirement defined in the current Laboratory Manual.

* At least 1 lesion, not previously irradiated, not biopsied during the screening period, that can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes which must have short axis ≥15 mm) with CT or MRI which is suitable for accurate repeated measurements. If only 1 measurable lesion exists, it is acceptable to be used as long as baseline tumour assessment scans are done at least 14 days after the screening tumour sample collection is performed.
* Prior lines of therapy in locally advanced/metastatic setting: Only prior 1L osimertinib treatment in metastatic setting is permitted.
* Adequate haematological function defined as:
* Absolute neutrophil count ≥1500/μL
* Haemoglobin ≥9 g/dL (no transfusion in the past 2 weeks)
* Platelets ≥100,000/μL (no transfusion in the past 10 days)
* Adequate liver function
* ALT, AST ≤2.5 x ULN with TBL ≤ ULN OR
* TBL >ULN to ≤1.5x ULN with ALT and AST ≤ ULN
* Adequate renal function - defined as a serum creatinine <1.5 times the institutional ULN OR a glomerular filtration rate ≥50 mL/min. Confirmation of creatinine clearance is only required when creatinine is only required when creatinine is >1.5 times ULN.
* Adequate coagulation parameters: INR <1.5 and activated partial thromboplastin time <1.5 x ULN unless patients are receiving therapeutic anti coagulation which affects these parameters.
* Patients with known tumour thrombus or deep vein thrombosis are eligible if clinically stable on low molecular weight heparin for ≥2 weeks. The use of direct oral anticoagulants such as apixaban/rivaroxaban will be accepted as treatment for cancer related thromboembolism treatment. The use of warfarin for oral anticoagulation is not recommended.
* ECOG/WHO performance status of 0 or 1 with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks.
* Females must be using highly effective contraceptive measures, should not be breast feeding and must have a negative pregnancy test if of childbearing potential, or must have evidence of non-childbearing potential.
* Males with a female partner of childbearing potential should be willing to use barrier contraception during the study and for 6 months following discontinuation of study drug.

Exclusion Criteria:

* Unresolved toxicities from any prior therapy greater than CTCAE Grade 1 at the time of starting study treatment with the exception of alopecia and Grade 2 prior platinum therapy related neuropathy.
* As judged by the investigator, active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of oral therapy (eg, ulcerative disease, uncontrolled nausea, vomiting, diarrhoea Grade ≥2, malabsorption syndrome or previous significant bowel resection).
* Any of the following cardiac diseases currently or within the last 6 months:

Unstable angina pectoris

Congestive heart failure (New York Heart Association [NYHA] ≥Grade 2)

Acute myocardial infarction

Stroke or transient ischemic attack

Uncontrolled hypertension (blood pressure [BP] ≥150/95 mmHg despite medical therapy).

Mean resting correct QT interval (QTcF) >470 msec for women and >450 msec for men at Screening, obtained from 3 ECGs using the screening clinic ECG machine derived QTcF value.

Any factors that may increase the risk of QTcF prolongation or risk of arrhythmic events such as heart failure, chronic hypokalaemia not correctable with supplements, congenital or familial long QT syndrome, family history of unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval and cause Torsade de Pointes.

Any clinically important abnormalities in rhythm, conduction or morphology of resting ECGs, eg, complete left bundle branch block, third degree heart block, second degree heart block, P-R interval >250 msec.

Acute coronary syndrome

* Wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) administered ≤28 days or limited field radiation for palliation ≤7 days prior to starting study drug or has not recovered from side effects of such therapy.
* Major surgical procedures ≤28 days of beginning study drug or minor surgical procedures ≤7 days
* Evidence of severe or uncontrolled systemic diseases, including renal transplant, active bleeding diatheses or uncontrolled hypertension, which in the investigator's opinion makes it undesirable for the patient to participate
* Active hepatitis B or C or known serious active infection e.g. tuberculosis or human immunodeficiency virus. Viral testing is not required for assessment of eligibility for the study.
* Known serious active infection including, but not limited to, tuberculosis, or human immunodeficiency virus (positive human immunodeficiency virus 1/2 antibodies).
* Presence of other active cancers, or history of treatment for invasive cancer, within the last 5 years. Patients with Stage I cancer who have received definitive local treatment at least 3 years previously, and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma (ie, non-invasive) are eligible, as are patients with history of non-melanoma skin cancer.
* Spinal cord compression or brain metastases unless asymptomatic, stable and not requiring steroids for at least 2 weeks prior to start of study treatment.
* Past medical history of interstitial lung disease(ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
* History of liver cirrhosis of any origin and clinical stage; or history of other serious liver disease or chronic disease with relevant liver involvement, with or without normal LFTs,
* Prior or current treatment with a 3rd generation EGFR-TKI other than osimertinib
* Prior or current treatment with savolitinib or another MET inhibitor (eg, foretinib, crizotinib, cabozantinib, onartuzumab, capmatinib).
* Any cytotoxic chemotherapy, investigational agents or other anticancer drugs for the treatment of advanced NSCLC from a previous treatment regimen or clinical study within 14 days prior to the first dose of study treatment with the exception of monotherapy osimertinib which may continue uninterrupted during screening.
* Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers of CYP3A4, strong inhibitors of CYP1A2 within 3 weeks of the first dose of study treatment (including St John's Wort).
* Participation in another clinical study with a cytotoxic, investigational product (IP), or other anticancer drug for the treatment of advanced NSCLC if received IP from that study within 14 days of the first dose of study treatment.
* Known hypersensitivity to the active or inactive excipients of osimertinib or savolitinib or drugs with a similar chemical structure or class.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lecia V Sequist, MD MPH, Principal Investigator — Massachusetts General Hospital; Myung-Ju Ahn, MD, Principal Investigator — Samsung Medical Centre Sungkyunkwan University School of Medicine
Locations (77):
- United States (11):
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, Sacramento, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Rochester, Minnesota
  - Research Site, Brooklyn, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Seattle, Washington
- Brazil (8):
  - Research Site, Barretos
  - Research Site, Curitiba
  - Research Site, Goiânia
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Canada (5):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Newmarket, Ontario
  - Research Site, North York, Ontario
  - Research Site, Toronto, Ontario
- Research Site, Santiago, Chile
- Denmark (6):
  - Research Site, Aalborg
  - Research Site, Herlev
  - Research Site, København Ø
  - Research Site, Næstved
  - Research Site, Odense
  - Research Site, Vejle
- France (5):
  - Research Site, Dijon
  - Research Site, Marseille
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Rennes
- India (4):
  - Research Site, Bangalore
  - Research Site, Chennai
  - Research Site, Kolkata
  - Research Site, New Delhi
- Italy (8):
  - Research Site, Avellino
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Orbassano
  - Research Site, Padua
  - Research Site, Parma
  - Research Site, Perugia
  - Research Site, Peschiera del Garda
- Japan (10):
  - Research Site, Fukuoka
  - Research Site, Hiroshima
  - Research Site, Kanazawa
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Sapporo
  - Research Site, Sayama
  - Research Site, Sunto-gun
  - Research Site, Wakayama
  - Research Site, Yokohama
- South Korea (4):
  - Research Site, Goyang-si
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (6):
  - Research Site, Córdoba
  - Research Site, Donostia / San Sebastian
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Valencia
  - Research Site, Zaragoza
- Taiwan (7):
  - Research Site, Hsinchu
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Vietnam (2):
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Yang JC, Chen YM, Batra U, Do KH, Sitthideatphaiboon P, Danchaivijitr P, Lee KY, Chindaprasirt J, Yang CT, Chang GC, Charoentum C, Ungtrakul T, Moran JIH, Hartmaier R, Igwegbe I, Gont A, Haskins M, Xu W, Riess JW. Savolitinib Plus Osimertinib in Epidermal Growth Factor-Mutated, MET-Amplified Advanced Non-Small Cell Lung Cancer: A Randomized Phase II trial. Clin Lung Cancer. 2025 Oct 22;27(1):38-46. doi: 10.1016/j.cllc.2025.10.018. Online ahead of print. PMID 41308232
- [Derived] Schmid S, Fruh M, Peters S. Targeting MET in EGFR resistance in non-small-cell lung cancer-ready for daily practice? Lancet Oncol. 2020 Mar;21(3):320-322. doi: 10.1016/S1470-2045(19)30859-9. Epub 2020 Feb 3. No abstract available. PMID 32027845
- See also: Redacted Statistical Analysis Plan (SAP) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5084C00007&attachmentIdentifier=a25a99af-a8aa-403a-8745-71929862fc7a&fileName=D5084C00007_-___Statistical_Analysis_Plan_for_redaction_MH_Redacted.pdf&versionIdentifier=
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5084C00007&attachmentIdentifier=35897367-5cc1-4164-933d-fef87459aec6&fileName=d5084c00007-study-synopsis_for_redaction_Redacted.pdf&versionIdentifier=
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5084C00007&attachmentIdentifier=7e52c879-6716-4e4b-a8a0-bae62baa9450&fileName=d5084c00007-csp-v8-redacted_(1).pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the study involved prescreening with central FISH/IHC for MET amplification/overexpression. Eligible participants (FISH5+/IHC50+ for CSP v1.0-v6.0; FISH10+/IHC90+ for CSP v7.0) proceeded to screening for full eligibility. After screening, assignment or randomization to a treatment cohort depended on the applicable CSP version.
Pre-assignment Details: One site inadvertently processed a dosing transaction in IxRS causing the PRF enrollment number (367) to be higher than the enrollment number in the PRF (366).
Groups:
- Savo 300mg QD + Osi: All patients assigned to savolitinib 300 mg qd + osimertinib and who received >=1 dose of either study treatment.
- Savo 300mg BID + Osi: All patients assigned to savolitinib 300 mg bid + osimertinib and who received >=1 dose of either study treatment.
- Savo 600mg QD + Osi: All patients assigned to savolitinib 600 mg qd + osimertinib and who received >=1 dose of either study treatment.
- Savo 300mg BID Monotherapy: All patients assigned to savolitinib 300 mg bid + placebo and who received >=1 dose of either study treatment.
Period: Overall Study
Arm/Group | Savo 300mg QD + Osi | Savo 300mg BID + Osi | Savo 600mg QD + Osi | Savo 300mg BID Monotherapy
Started | 196 | 101 | 44 | 25
Completed (All patients remain on study or in survival follow-up until death or withdrawl of consent.) | 0 | 0 | 0 | 0
Not Completed | 196 | 101 | 44 | 25
Not completed — Death | 163 | 68 | 36 | 9
Not completed — Withdrawal by Subject | 19 | 1 | 5 | 2
Not completed — Ongoing on-study | 14 | 32 | 3 | 13
Not completed — Incorrectly Randomized | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Patients assigned to study treatment and receiving >=1 dose of study treatment.
Groups:
- 300 mg QD + Osi: All patients assigned to savolitinib 300 mg qd + osimertinib and who have received >=1 dose of either study drug.
- Savo 300 mg BID + Osi: All patients assigned to savolitinib 300 mg bid + osimertinib and who received >=1 dose of either study treatment.
- 600 mg QD + Osi: All patients assigned to savolitinib 600 mg qd + osimertinib and who received >=1 dose of either study treatment.
- Total: Total of all reporting groups
Arm/Group | 300 mg QD + Osi | Savo 300 mg BID + Osi | 600 mg QD + Osi | Savo 300mg BID Monotherapy | Total
Number analyzed (Participants) | 196 | 101 | 44 | 24 | 365
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.5 (11.27) | 63.4 (10.89) | 62.0 (12.14) | 65.0 (10.64) | 62.3 (11.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 29 | 23 | 9 | 135
  Male | 122 | 72 | 21 | 15 | 230
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 105 | 31 | 22 | 12 | 170
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 3 | 0 | 4
  White | 77 | 66 | 18 | 12 | 173
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 13 | 3 | 1 | 0 | 17
Region of Enrollment [Number; unit: Participants]
  Brazil | 13 | 2 | 1 | 0 | 16
  CAN | 13 | 16 | 6 | 7 | 42
  Chile | 6 | 0 | 0 | 0 | 6
  Denmark | 6 | 2 | 0 | 1 | 9
  Spain | 3 | 3 | 3 | 1 | 10
  France | 10 | 2 | 1 | 0 | 13
  India | 6 | 1 | 1 | 1 | 9
  Italy | 39 | 47 | 14 | 5 | 105
  Japan | 18 | 0 | 0 | 0 | 18
  Korea, Republic Of | 47 | 7 | 16 | 4 | 74
  Taiwan, China | 7 | 12 | 2 | 3 | 24
  USA | 21 | 9 | 0 | 2 | 32
  Viet Nam | 7 | 0 | 0 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) by Investigator Assessment; Target Population Analysis Set
Description: Percentage of subjects with a confirmed Objective Response (OR) per Response Evaluation Criteria In Solid Tumors (RECIST 1.1). OR includes Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: ≥30% decrease in target lesion diameters). OR must be recorded at one visit and confirmed by repeat imaging at least 4 weeks later, with no disease progression between initial and confirmation visits.
Time Frame: Time from randomization/first dose of study treatment to progression or last evaluable assessment in the absence of progressionuntil the end of the study, or an approximate maximum of 5.6 years.
Population: All patients assigned to savolitinib 300 mg bid + osimertinib with EGFRm+ and MET amplified/overexpressed (FISH10+ and/or IHC90+), locally advanced or metastatic NSCLC who have progressed following treatment with 1L osimertinib, and have taken >=1 dose of either study drug.
Measure: Number (95% Confidence Interval); unit: Percent of subjects
Arm/Group | Savo 300 mg BID + Osi
Number analyzed (Participants) | 80
Percent of subjects | 56.3 [44.70 to 67.32]

2. Primary Outcome: Objective Response Rate (ORR) by Investigator Assessment; 300 mg QD Safety Analysis Set
Description: as for outcome 1
Time Frame: Time from randomization/first dose of study treatment to progression or last evaluable assessment in the absence of progression until the end of the study, or an approximate maximum of 5.6 years.
Population: All enrolled patients who received ≥1 dose of either study drug.
Measure: Number (95% Confidence Interval); unit: Percent of subjects
Groups:
- Savo 300 mg QD + Osi: All patients assigned to savolitinib 300 mg QD + osimertinib and who received >=1 dose of either study drug.
Arm/Group | Savo 300 mg QD + Osi
Number analyzed (Participants) | 196
Percent of subjects | 31.6 [25.19 to 38.64]

3. Secondary Outcome: Objective Response Rate (ORR) by BICR Assessment; Target Population Analysis Set
Description: as for outcome 1
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percent of subjects
Arm/Group | Savo 300 mg BID + Osi
Number analyzed (Participants) | 80
Percent of subjects | 55.0 [43.5 to 66.2]

4. Secondary Outcome: Duration of Response (DoR) by Investigator Assessment; Target Population Analysis Set
Description: Median time of response for patients with an investigator assessed confirmed objective response per RECIST1.1
Time Frame: From date of first confirmed objective response to progressive disease in accordance with RECIST1.1 or death from any cause, whichever came first; assessed for up to 5.6 years.
Population: All patients with an objective response and assigned to savolitinib 300 mg bid + osimertinib who have FISH10+ and/or IHC90+ status, have progressed following 1L osimertinib, and have taken >=1 dose of either study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Savo 300 mg BID + Osi
Number analyzed (Participants) | 45
Months | 7.13 [5.55 to 9.63]

5. Secondary Outcome: Duration of Response (DoR) by BICR Assessment; Target Population Analysis Set
Description: Median time of response for patients with an investigator assessed confirmed objective response per RECIST1.1
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Savo 300 mg BID + Osi
Number analyzed (Participants) | 44
Months | 9.92 [6.01 to 13.73]

6. Secondary Outcome: Progression-free Survival (PFS) by Investigator Assessment; Target Population Analysis Set
Description: Median progression-free survival (PFS) was measured by investigator assessment using RECIST 1.1 and the Kaplan-Meier method. Progressive disease (PD) per RECIST 1.1 is defined as at least a 20% increase in the sum of target lesion diameters (with an absolute increase of ≥5 mm); unequivocal progression of non-target lesions, which may result from marked progression in a single lesion or multiple lesions; or the appearance of one or more unequivocal new lesions.
Time Frame: Time from randomization/start of study treatment to investigator assess progressive disease per RECIST1.1 or death, assessed for up to 5.6 years.
Population: All patients assigned to savolitinib 300 mg bid + osimertinib who have FISH10+ and/or IHC90+ status, have progressed following 1L osimertinib, and have taken >=1 dose of either study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Savo 300 mg BID + Osi
Number analyzed (Participants) | 80
Months | 7.39 [5.49 to 7.62]

7. Secondary Outcome: Progression-free Survival (PFS) by BICR Assessment; Target Population Analysis Set
Description: Median progression-free survival (PFS) was measured by BICR assessment using RECIST 1.1 and the Kaplan-Meier method. Progressive disease (PD) per RECIST 1.1 is defined as at least a 20% increase in the sum of target lesion diameters (with an absolute increase of ≥5 mm); unequivocal progression of non-target lesions, which may result from marked progression in a single lesion or multiple lesions; or the appearance of one or more unequivocal new lesions.
Time Frame: Time from randomization/start of study treatment to BICR assessed progressive disease per RECIST1.1 or death, assessed for up to 5.6 years.
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Savo 300 mg BID + Osi
Number analyzed (Participants) | 80
Months | 7.52 [6.37 to 11.33]

8. Secondary Outcome: Overall Survival (OS); Target Population Analysis Set
Description: Overall Survival (OS) from all-cause mortality
Time Frame: Time from randomization/start of study treatment to all-cause death, assessed for up to 5.6 years.
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Savo 300 mg BID + Osi
Number analyzed (Participants) | 80
Months | 14.42 [11.89 to 17.87]

9. Secondary Outcome: Objective Response Rate (ORR) by Investigator Assessment; Contribution of Components Analysis Set
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All patients randomized under CSP version 7.0 with treatment groups assigned in accordance with the randomization, regardless of the treatment actually received.
Measure: Number (95% Confidence Interval); unit: Percent of subjects
Groups:
- Savo 300 mg BID + Osi: All patients randomized to savolitinib 300 mg bid + osimertinib.
- Savo 300 mg BID Monotherapy: All patients randomized to savolitinib 300 mg bid + placebo.
Arm/Group | Savo 300 mg BID + Osi | Savo 300 mg BID Monotherapy
Number analyzed (Participants) | 48 | 25
Percent of subjects | 54.2 [39.2 to 68.6] | 24.0 [9.4 to 45.1]

10. Secondary Outcome: Objective Response Rate (ORR) by BICR Assessment; Contribution of Components Analysis Set
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percent of subjects
Arm/Group | Savo 300 mg BID + Osi | Savo 300 mg BID Monotherapy
Number analyzed (Participants) | 48 | 25
Percent of subjects | 58.3 [43.2 to 72.4] | 16.0 [4.5 to 36.1]

11. Secondary Outcome: Duration of Response (DoR) by Investigator Assessment; Contribution of Components Analysis Set
Description: Median time of response for patients with an investigator assessed confirmed objective response per RECIST1.1
Time Frame: as for outcome 4
Population: All patients with an objective response and randomized under CSP version 7.0 with treatment groups assigned in accordance with the randomization, regardless of the treatment actually received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Savo 300 mg BID + Osi | Savo 300 mg BID Monotherapy
Number analyzed (Participants) | 26 | 6
Months | 7.95 [4.90 to 11.73] | 4.71 [2.56 to NA] — The 95% CI upper limit of median PFS was not estimable at this analysis due to insufficient number of participants with events.

12. Secondary Outcome: Duration of Response (DoR) by BICR Assessment; Contribution of Components Analysis Set
Description: Median time of response for patients with an investigator assessed confirmed objective response per RECIST1.1
Time Frame: as for outcome 4
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Savo 300 mg BID + Osi | Savo 300 mg BID Monotherapy
Number analyzed (Participants) | 28 | 4
Months | 11.76 [6.01 to NA] — The 95% CI upper limit of median PFS was not estimable at this analysis due to insufficient number of participants with events. | 4.53 [2.56 to NA] — The 95% CI upper limit of median PFS was not estimable at this analysis due to insufficient number of participants with events.

13. Secondary Outcome: Progression-free Survival (PFS) by Investigator Assessment; Contribution of Components Analysis Set
Description: as for outcome 6
Time Frame: as for outcome 6
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Savo 300 mg BID + Osi | Savo 300 mg BID Monotherapy
Number analyzed (Participants) | 48 | 25
Months | 7.56 [5.55 to 11.04] | 2.66 [1.41 to 4.11]

14. Secondary Outcome: Progression-free Survival (PFS) by BICR Assessment; Contribution of Components Analysis Set
Description: as for outcome 7
Time Frame: as for outcome 7
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Savo 300 mg BID + Osi | Savo 300 mg BID Monotherapy
Number analyzed (Participants) | 48 | 25
Months | 8.28 [5.82 to 15.08] | 3.65 [1.41 to 5.75]

15. Secondary Outcome: Objective Response Rate (ORR) by Investigator Assessment; Safety Analysis Set
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All enrolled patients who take ≥1 dose of either study drug.
Measure: Number (95% Confidence Interval); unit: Percent of subjects
Groups:
- 300 mg BID + Osi: All patients assigned to savolitinib 300 mg bid + osimertinib and who received >=1 dose of either study treatment.
- Savo 600 mg QD + Osi: All patients assigned to savolitinib 600 mg qd + osimertinib and who have taken >=1 dose of either study drug.
Arm/Group | 300 mg BID + Osi | Savo 600 mg QD + Osi
Number analyzed (Participants) | 101 | 44
Percent of subjects | 51.5 [41.3 to 61.6] | 31.8 [18.6 to 47.6]

16. Secondary Outcome: Objective Response Rate (ORR) by BICR Assessment; Safety Analysis Set
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All enrolled patients who take ≥1 dose of either study drug.
Measure: Number (95% Confidence Interval); unit: Percent of subjects
Groups:
- Savo 600 mg QD + Osi: All patients assigned to savolitinib 600 mg qd + osimertinib and who have received >=1 dose of either study drug.
Arm/Group | 300 mg QD + Osi | 300 mg BID + Osi | Savo 600 mg QD + Osi
Number analyzed (Participants) | 196 | 101 | 44
Percent of subjects | 32.7 [26.1 to 39.7] | 49.5 [39.4 to 59.6] | 34.1 [20.5 to 49.9]

17. Secondary Outcome: Duration of Response (DoR) by Investigator Assessment; Safety Analysis Set
Description: Median time of response for patients with an investigator assessed confirmed objective response per RECIST1.1
Time Frame: as for outcome 4
Population: All enrolled patients with an objective response and who take ≥1 dose of either study drug.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Savo 300 mg QD + Osi: All patients assigned to savolitinib 300 mg qd + osimertinib and who received >=1 dose of either study treatment
- Savo 600 mg QD + Osi: All patients assigned to savolitinib 600 mg qd + osimertinib and who received >=1 dose of either study treatment
Arm/Group | Savo 300 mg QD + Osi | Savo 300 mg BID + Osi | Savo 600 mg QD + Osi
Number analyzed (Participants) | 62 | 52 | 14
Months | 8.54 [7.56 to 10.51] | 6.01 [4.90 to 9.07] | 8.59 [3.94 to 21.95]

18. Secondary Outcome: Duration of Response (DoR) by BICR Assessment; Safety Analysis Set
Description: Median time of response for patients with an investigator assessed confirmed objective response per RECIST1.1
Time Frame: as for outcome 4
Population: All enrolled patients who take ≥1 dose of either study drug and with an objective response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Savo 300 mg QD + Osi | Savo 300 mg BID + Osi | Savo 600 mg QD + Osi
Number analyzed (Participants) | 64 | 50 | 15
Months | 9.66 [7.49 to 13.17] | 9.92 [6.11 to 12.42] | 18.86 [7.72 to 24.67]

19. Secondary Outcome: Overall Survival (OS); Safety Analysis Set
Description: Overall Survival (OS) from all-cause mortality
Time Frame: Time from randomization/start of study treatment to all-cause death, assessed for up to 5.6 years.
Population: All enrolled patients who take ≥1 dose of either study drug
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Savo 300 QD + Osi: All patients assigned to savolitinib 300 mg qd + osimertinib and who received >=1 dose of either study treatment.
Arm/Group | Savo 300 QD + Osi | Savo 300 mg BID + Osi | Savo 600 mg QD + Osi
Number analyzed (Participants) | 196 | 101 | 44
Months | 14.75 [12.88 to 17.02] | 13.90 [11.76 to 15.87] | 15.08 [9.17 to 18.60]

20. Secondary Outcome: Progression-free Survival (PFS) by Investigator Assessment; Safety Analysis Set
Description: as for outcome 6
Time Frame: as for outcome 6
Population: All enrolled patients who take ≥1 dose of either study drug.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Savo 600 mg QD + Osi: All patients assigned to savolitinib 600 mg qd + placebo and who received >=1 dose of either study treatment.
Arm/Group | Savo 300 QD + Osi | Savo 300 mg BID + Osi | Savo 600 mg QD + Osi
Number analyzed (Participants) | 196 | 101 | 44
Months | 5.29 [4.17 to 5.78] | 5.68 [4.27 to 7.39] | 4.40 [2.56 to 7.43]

21. Secondary Outcome: Progression-free Survival (PFS) by BICR Assessment; Safety Analysis Set
Description: as for outcome 7
Time Frame: as for outcome 7
Population: All enrolled patients who take ≥1 dose of either study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Savo 300 QD + Osi | Savo 300 mg BID + Osi | Savo 600 mg QD + Osi
Number analyzed (Participants) | 196 | 101 | 44
Months | 5.55 [4.86 to 7.36] | 7.39 [5.59 to 9.20] | 4.44 [2.53 to 9.33]

ADVERSE EVENTS:
Time Frame: AEs with an onset date or worsening on or after the first dose and up to and including 35 days after the last dose of study treatment, or prior to the initiation of crossover treatment, or start of subsequent anti-cancer therapy. Cross-over period includes AEs with an onset or worsening on or after start of crossover therapy and up to 35 days following the last dose of crossover treatment or start of subsequent anti-cancer therapy. Followed for a maximum of 5.6 years.
Groups:
- Cross-over: Includes all subjects randomized to Savolitinib 300 mg BID + placebo, who crossed over to Savolitinib 300 mg BID + Osimertinib 80 mg QD after disease progression.
Arm/Group | Savo 300mg QD + Osi | Savo 300mg BID + Osi | Savo 600mg QD + Osi | Savo 300mg BID Monotherapy | Cross-over
All-Cause Mortality (participants affected / at risk) | 164/196 | 68/101 | 37/44 | 9/24 | 3/14
Serious Adverse Events (participants affected / at risk) | 62/196 | 31/101 | 20/44 | 8/24 | 1/14
Other Adverse Events (participants affected / at risk) | 185/196 | 99/101 | 42/44 | 22/24 | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Savo 300mg QD + Osi (N=196) | Savo 300mg BID + Osi (N=101) | Savo 600mg QD + Osi (N=44) | Savo 300mg BID Monotherapy (N=24) | Cross-over (N=14)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inner ear disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transurethral bladder resection (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperpyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Colonic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extradural abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 4 (5) | 3 (4) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis chemical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sars-cov-2 test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Savo 300mg QD + Osi (N=196) | Savo 300mg BID + Osi (N=101) | Savo 600mg QD + Osi (N=44) | Savo 300mg BID Monotherapy (N=24) | Cross-over (N=14)
Dizziness (Nervous system disorders) | 17 (19) | 9 (12) | 6 (6) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 22 (31) | 9 (11) | 3 (3) | 1 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 3 (3) | 3 (3) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 14 (14) | 5 (5) | 3 (3) | 0 (0) | 2 (2)
Dysuria (Renal and urinary disorders) | 7 (8) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 26 (29) | 15 (17) | 6 (7) | 4 (4) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30 (33) | 19 (22) | 8 (12) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 1 (1) | 6 (8) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 10 (10) | 5 (5) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 10 (11) | 5 (5) | 5 (6) | 3 (3) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 10 (13) | 4 (8) | 1 (1) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 12 (16) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 19 (22) | 12 (15) | 6 (6) | 2 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 25 (27) | 12 (18) | 7 (8) | 2 (2) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 6 (6) | 8 (8) | 7 (7) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 2 (2) | 7 (7) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 7 (7) | 7 (7) | 3 (4) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 10 (11) | 9 (11) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 30 (34) | 15 (15) | 9 (11) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 35 (56) | 33 (52) | 11 (19) | 2 (2) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 18 (23) | 8 (8) | 9 (10) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (5) | 5 (5) | 1 (1) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 77 (91) | 45 (61) | 15 (19) | 5 (6) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 9 (17) | 6 (7) | 2 (2) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 38 (65) | 21 (37) | 12 (17) | 3 (3) | 0 (0)
Asthenia (General disorders) | 20 (21) | 19 (21) | 4 (4) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 7 (11) | 7 (7) | 4 (5) | 0 (0) | 0 (0)
Chills (General disorders) | 5 (5) | 1 (2) | 3 (5) | 1 (1) | 0 (0)
Fatigue (General disorders) | 38 (42) | 17 (19) | 9 (10) | 4 (4) | 1 (1)
Oedema peripheral (General disorders) | 79 (108) | 59 (91) | 19 (28) | 10 (15) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (6) | 9 (9) | 1 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 25 (27) | 18 (24) | 11 (12) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 6 (6) | 12 (13) | 3 (3) | 1 (1) | 2 (2)
Paronychia (Infections and infestations) | 37 (47) | 14 (17) | 7 (9) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 6 (6) | 6 (8) | 2 (2) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (10) | 6 (8) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 8 (9) | 12 (14) | 4 (4) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 13 (16) | 10 (12) | 7 (11) | 1 (1) | 1 (1)
Amylase increased (Investigations) | 9 (9) | 11 (16) | 3 (5) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 14 (21) | 6 (8) | 6 (10) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 7 (7) | 7 (7) | 5 (5) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 11 (15) | 6 (7) | 4 (6) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 12 (19) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Platelet count decreased (Investigations) | 7 (9) | 6 (11) | 4 (5) | 2 (3) | 0 (0)
Weight decreased (Investigations) | 7 (7) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 10 (14) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 41 (44) | 13 (14) | 12 (13) | 3 (3) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 17 (19) | 15 (26) | 3 (7) | 2 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 16 (19) | 10 (11) | 5 (10) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (8) | 8 (8) | 2 (2) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 8 (10) | 2 (2) | 2 (3) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 (30) | 12 (13) | 5 (5) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (13) | 15 (16) | 7 (7) | 2 (2) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 (13) | 7 (7) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (20) | 5 (6) | 2 (2) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 (18) | 11 (15) | 5 (7) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
No limitations or caveats were identified in this analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-05-24): https://cdn.clinicaltrials.gov/large-docs/29/NCT03778229/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT03778229/SAP_001.pdf